CLINICAL TRIAL: NCT06310733
Title: The Effects of Probiotics, Lactobacillus GG, in the Treatment of Abdominal Pain in Children With Functional Abdominal Pain Disorders - A Randomized Controlled Trial
Brief Title: The Effects of Probiotics, Lactobacillus GG, in the Treatment of Abdominal Pain in Children With Functional Abdominal Pain Disorders
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Atchariya Chanpong, Division of Gastroenterology and Hepatology, Department of Pediatrics, Faculty of Medicine, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC 66-517-1-1
Record Dates: First submitted 2024-02-26; First posted 2024-03-15 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Functional Abdominal Pain Syndrome
Keywords: Functional Abdominal Pain Syndrome; Brain-Gut-Microbiome Axis; microbiome; irritable bowel syndrome; microbiota
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LGG (ATCC 53103) (Experimental): A suspension of freeze-dried LGG ATCC53103 in excipients in an aqueous solution supplied in a 10-mL dark bottle with a delivery cap.
  Interventions: Drug: LGG
- Placebo (Placebo Comparator): An identical aqueous solution in appearance and taste but without LGG.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LGG — Participants will take 10 mL of a suspension of freeze-dried LGG ATCC53103 in excipients in an aqueous solution, supplied in a 10-mL dark bottle with a delivery cap.
  Arms: LGG (ATCC 53103)
Drug: Placebo — Participants will take 10 mL of an identical aqueous solution in appearance and taste but without LGG, supplied in a 10-mL dark bottle.
  Arms: Placebo

SUMMARY:
Recurrent or chronic abdominal pain is one of the common gastrointestinal problems in children. While most children do not have organic origins (so called functional abdominal pain disorders; FAPDs), the symptoms can nevertheless be severe enough to impair the patient's quality of life, growth, and development. To help rule out organic disorders and diagnose this condition, some individuals underwent multiple invasive and costly studies.

Generally, the diagnosis of FAPDs is based on clinical symptoms and criteria, it can be divided into irritable bowel syndrome (IBS), abdominal migraine, functional abdominal pain (FAP) and functional dyspepsia (FD). Approximately 14% of children globally, between the ages of 4 and 18, experience functional abdominal pain issues8. In Thailand, the prevalence of FAPDs among adolescents (mean age of 16 years) was 5.3%, functional dyspepsia and irritable bowel syndrome were found to be the most prevalent subtypes.

The pathogenesis of FAPDs is believed to result from disruptions in the microbiota-gut-brain axis, which may happen early in life or throughout. Hence, several studies, specifically in western countries, reported the role of probiotics, specifically Lactobacillus rhamnosus GG (LGG), in modulating abdominal symptoms in children with FAPDs.

It is widely known that the diversity of gut microbiota depends on multiple factors including ethnicity, mode of delivery, dietary and environmental factors. However, the studies on the use of probiotics in pediatric patients with FAPDs have been mainly conducted in western countries. Since there are limited studies on the effectiveness of probiotics in Asian children with FAPDs, the investigators aim to evaluate the effects of probiotics, LGG, in the treatment of children who suffered from FAPDs.

The secondary objectives are to measure daily pain score in children with and without FAPDs, to evaluate and compare the diversity of fecal microbiota in children with FAPDs and those without FAPDs, and to compare the diversity of fecal microbiota between children with FAPDs who took probiotics and those who did not.

ELIGIBILITY:
Inclusion Criteria:

* Children, aged 6-15 years old, with a diagnosis of IBS or FAP, according to the Rome IV diagnostic criteria. The diagnosis of IBS or FAP was based on a clinical interview performed by pediatric gastroenterologist.

For healthy controls: non-obese children, aged 6-15 years old, without any gastrointestinal symptoms at the time of recruitment.

Exclusion Criteria:

* Children who

  1. had any chronic diseases, including neurobehavioral disorders
  2. received treatment with antibiotics/probiotics in the previous 2 months
  3. received medication that affects gastrointestinal motility in the previous 1 week
  4. had a pain history suggestive of functional dyspepsia/aerophagia/abdominal migraine/functional constipation
  5. exhibited growth failure
  6. had gastrointestinal obstructions/stricture
  7. displayed alarming signs of organic condition
  8. had previous abdominal surgery
  9. had abnormal baseline test results as part of their standard work-up (e.g. complete blood counts; erythrocyte sedimentation rate; liver-pancreas-kidney function tests; stool examination for occult blood, ova, and parasites; fecal calprotectin; urinalysis; abdominal ultrasound; 13C-urea breath test; gastric emptying study, if any)
  10. had family history of peptic ulcer disease or inflammatory bowel disease

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 54 (Estimated)
Dates: Start 2024-03-21 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
The response rate of 4 week-probiotics (LGG) on the severity of abdominal pain (number of episodes or the intensity of pain), compared to the conventional treatment, in children who suffered from FAPDs | 12 weeks
  Faces pain scale (0-6); higher scores mean a worse outcome.
The response rate of 4 week-probiotics (LGG) on the severity of abdominal pain (number of episodes or the intensity of pain), compared to the conventional treatment, in children who suffered from FAPDs | 12 weeks
  Visual analog scale (0-10); higher scores mean a worse outcome.
The response rate of 4 week-probiotics (LGG) on the severity of abdominal pain (number of episodes or the intensity of pain), compared to the conventional treatment, in children who suffered from FAPDs | 12 weeks
  Daily food and symptom record

SECONDARY OUTCOMES:
To measure daily pain score in children with and without FAPDs | 12 weeks
  Faces pain scale (0-6); higher scores mean a worse outcome.
To measure daily pain score in children with and without FAPDs | 12 weeks
  Visual analog scale (0-10); higher scores mean a worse outcome.
To measure daily pain score in children with and without FAPDs | 12 weeks
  Daily food and symptom record
To compare the diversity of fecal microbiota in children with FAPDs who took probiotics and those who did not | 4 weeks
  stool samples for rDNA sequencing before and after 4 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Atchariya Chanpong, Songkhla, Thailand